CLINICAL TRIAL: NCT01874119
Title: Phase 2B Double Blind Placebo Controlled Crossover Study Evaluating the Efficacy of IV Fosaprepitant for Chemo Induced N/V With High Dose Interleukin 2 for Metastatic Melanoma and Metastatic Renal Cell Carcinoma
Brief Title: Fosaprepitant for N/V With High-dose Interleukin-2 for Metastatic Melanoma and Renal Cell Carcinoma
Acronym: HDIL2/Emend
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment issues
Sponsor: St. Louis University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, John Richart, M.D., Associate Professor, Dept. of Internal Medicine, Hematology and Oncology, St. Louis University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Merck-MISP-50440, 23432
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: melanoma; renal cell carcinoma; interleukin-2
MeSH Terms: conditions — Vomiting; Melanoma; Carcinoma, Renal Cell | interventions — fosaprepitant; Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fosaprepitant (Experimental): During treatment admission, intravenous fosaprepitant 150 mg every 48 hours during 6-day hospital admission
  Interventions: Drug: Fosaprepitant
- Placebo (Placebo Comparator): During placebo admission, intravenous 0.9% saline every 48 hours during 6-day hospital admission
  Interventions: Drug: Fosaprepitant

INTERVENTIONS:
Drug: Fosaprepitant — During treatment admission, intravenous fosaprepitant 150 mg every 48 hours during 6-day hospital admission
  Other Names: Emend

SUMMARY:
The purpose of this study is to investigate the effectiveness of intravenous fosaprepitant therapy to reduce nausea and vomiting during the treatment of high dose interleukin-2 (HD IL-2) therapy for metastatic melanoma or metastatic renal cell carcinoma. Fosaprepitant is an intravenous (IV) medication that is FDA- approved for use in adults for the prevention of nausea and vomiting during chemotherapy. Fosaprepitant works by blocking the neurokinin-1 receptor, which is a receptor in the brain that is known to cause nausea and vomiting. Past studies estimate that up to 70% of patients undergoing treatment with HD IL-2 will have nausea and/or vomiting. While fosaprepitant has been used in clinical practice to treat nausea and vomiting during HD IL-2, there have not been any studies done to see how well it works. All patients will receive treatment (IV fosaprepitant) during the study during either the first or second hospital admission for HD IL-2. On the admission that the subject is not receiving IV fosaprepitant, the subject will receive placebo (a medicine that looks like fosaprepitant, but is not active). The study is double-blinded, which means neither the subject, nor the study doctor will know to which group you have been assigned to that admission (IV fosaprepitant or placebo). This study design was chosen to limit the potential for bias, which means the trial was designed to try to ensure that unknown factors do not affect trial results. When patients start the study, patients will be randomly assigned to one of two groups: those who receive treatment (IV fosaprepitant) first and those who receive placebo first. During the first admission, subjects will be given the IV fosaprepitant or IV placebo during admission. During the second admission, subjects will 'crossover' and receive the other treatment that they did not receive during the first admission. Improvement in nausea and vomiting will be assessed by counting the number of nausea and vomiting episodes, recording if the subject needs additional medication for nausea and vomiting, and by using patient questionnaires.

DETAILED DESCRIPTION:
This is a Phase 2B double-blind placebo-controlled crossover study evaluating the efficacy of intravenous fosaprepitant for chemotherapy-induced nausea and vomiting in patients undergoing high-dose interleukin-2 (HD IL-2) therapy (720,000 IU/kg per dose intravenously; 14 doses, 2 cycles per course) for metastatic melanoma and metastatic renal cell carcinoma. A total of 22 subjects will be enrolled in the study. On study entry, patients will be randomized to receive either IV fosaprepitant (150 mg on Day 1, Day 3, or Day 5) or matched placebo during first admission of HD IL-2 therapy (cycle 1). All subjects will crossover and receive the opposite treatment during cycle 2. All patients will receive ondansetron 24 mg by mouth daily per standard protocol every 24 hours during Days 1-5 of admission starting 30 minutes prior to first dose of HD IL-2. During the treatment phase, subjects will receive Patients will receive IV fosaprepitant 30 minutes before first dose of HD IL-2 therapy and every 48 hours until completion of HD IL-2 therapy. Upon study entry, the subjects will be given a dairy to report episodes of vomiting, use of rescue therapy, and nausea assessments using the 1-100 scale within the visual analogue scale (VAS). The subject will be instructed to complete entries from baseline assessment (prior to first dose) until 5 days after last dose of HD IL-2 for endpoint analysis. During inpatient admissions, subjects will complete diary entries before each dose (q8 hours). As an outpatient, subjects will complete diary entries on a daily basis. Recording of whether or not pruritus was observed will also be collected within the subject diary. If a patient reports pruritus, the severity of pruritus on the 1-100 scale visual analogue scale (VAS) will also be collected. The study team will record any episodes of vomiting and the use of rescue therapy and ensure completion of patient diary during inpatient portion. Assessments will be made via telephone contact to determine onset of any episodes of CINV during outpatient portion. Safety assessments including adverse events (AEs) monitoring will be performed and assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

  1. Evidence of a personally signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial.
  2. Subjects who are willing to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
  3. Be at least 18 years of age at the time of informed consent.
  4. Has a diagnosis of metastatic melanoma or metastatic renal cell carcinoma and who will undergo high-dose interleukin-2 (HD IL-2) therapy
  5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less at Baseline/Day 1 visit. (See Appendix 6 on p. 51, ECOG Performance Status)
  6. Female of reproductive potential must agree use non-hormonal methods to avoid pregnancy during study participation and for 1 month after last dose of study drug

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the study:

  1. Women who are pregnant or lactating, or planning pregnancy
  2. Women of childbearing potential who refuse to use non-hormonal methods to avoid pregnancy
  3. Known hypersensitivity to any component of fosaprepitant or aprepitant
  4. Have taken pimozide or cisapride <4 weeks, cytochrome P450 3A4 inducers within 30 days, strong CYP3A4 inhibitors within 7 days, or antiemetics within 48 hours prior to treatment initiation (See Appendix 7 on p. 52 for list of CYP3A4 inducers and strong CYP3A4 inhibitors)
  5. Have evidence of clinically significant and unstable diseases or conditions such as cardiovascular, immunosuppressive, hematologic, hepatic, neurologic, renal, endocrine, collagen-vascular, or gastrointestinal abnormalities that the investigator thinks may interfere with study participation
  6. Participation in other study using an investigational or experimental therapy or procedure within 4 weeks or 5 half-lives (whichever is longer) before study entry
  7. Subjects cannot participate in studies of other investigational or experimental therapies or procedures at any time during their participation in this study.
  8. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
  9. Subjects who are investigational site staff members or who are Sponsor employees directly involved in the conduct of the trial.
  10. A subject who, in the opinion of the investigator or sponsor, will be uncooperative or unable to comply with study procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12-03 (Actual); Study Completion 2015-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Richart, M.D., Principal Investigator — Saint Louis University, Department of Internal Medicine, Division of Hematology and Oncology
Locations (1):
- Saint Louis University Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Grunberg S, Chua D, Maru A, Dinis J, DeVandry S, Boice JA, Hardwick JS, Beckford E, Taylor A, Carides A, Roila F, Herrstedt J. Single-dose fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting associated with cisplatin therapy: randomized, double-blind study protocol--EASE. J Clin Oncol. 2011 Apr 10;29(11):1495-501. doi: 10.1200/JCO.2010.31.7859. Epub 2011 Mar 7. PMID 21383291
- [Background] Van Laere K, De Hoon J, Bormans G, Koole M, Derdelinckx I, De Lepeleire I, Declercq R, Sanabria Bohorquez SM, Hamill T, Mozley PD, Tatosian D, Xie W, Liu Y, Liu F, Zappacosta P, Mahon C, Butterfield KL, Rosen LB, Murphy MG, Hargreaves RJ, Wagner JA, Shadle CR. Equivalent dynamic human brain NK1-receptor occupancy following single-dose i.v. fosaprepitant vs. oral aprepitant as assessed by PET imaging. Clin Pharmacol Ther. 2012 Aug;92(2):243-50. doi: 10.1038/clpt.2012.62. Epub 2012 Jun 27. PMID 22739139

RESULTS

PARTICIPANT FLOW:
Groups:
- Fosaprepitant First, Then Placebo: Fosaprepitant: During treatment admission, intravenous fosaprepitant 150 mg every 48 hours during 6-day hospital admission
  Placebo: During placebo admission, intravenous 0.9% saline every 48 hours during 6-day hospital admission
- Placebo First, Then Fosaprepitant: Placebo: During placebo admission, intravenous 0.9% saline every 48 hours during 6-day hospital admission
  Fosaprepitant: During treatment admission, intravenous fosaprepitant 150 mg every 48 hours during 6-day hospital admission
Period: First Intervention (6 Days)
Arm/Group | Fosaprepitant First, Then Placebo | Placebo First, Then Fosaprepitant
Started | 8 | 5
Completed | 7 | 5
Not Completed | 1 | 0
Period: Washout (7 Days)
Arm/Group | Fosaprepitant First, Then Placebo | Placebo First, Then Fosaprepitant
Started | 7 | 5
Completed | 4 | 3
Not Completed | 3 | 2
Period: Second Intervention (6 Days)
Arm/Group | Fosaprepitant First, Then Placebo | Placebo First, Then Fosaprepitant
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Participants Completing All Cycles: Fosaprepitant: During treatment admission, intravenous fosaprepitant 150 mg every 48 hours during 6-day hospital admission
  Placebo: intravenous 0.9% saline every 48 hours during 6-day hospital admission
Arm/Group | Study Participants Completing All Cycles
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 61 [37 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Response During Inpatient Admission
Description: No vomiting from the initiation of through 48 hours following the final dose of HD IL-2
Time Frame: From the initiation of through 48 hours following the final dose of Interleukin-2
Measure: Count of Participants; unit: Participants
Arm/Group | Fosaprepitant | Placebo
Number analyzed (Participants) | 7 | 7
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: From the initiation of through 48 hours following the final dose of HD IL-2
Arm/Group | Fosaprepitant | Placebo
All-Cause Mortality (participants affected / at risk) | 2/11 | 2/9
Serious Adverse Events (participants affected / at risk) | 3/11 | 4/9
Other Adverse Events (participants affected / at risk) | 11/11 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant (N=11) | Placebo (N=9)
Upper GI hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other - Uncal herniation (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Autoimmune disorder - Myocarditis (Immune system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant (N=11) | Placebo (N=9)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2) | 3 (3)
Platelet count decreased (Investigations) | 2 (2) | 1 (1)
Urine output decreased (Investigations) | 3 (3) | 4 (4)
Weight gain (Investigations) | 3 (3) | 3 (3)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbunemia (Metabolism and nutrition disorders) | 8 (8) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Cerebral edema (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Caution is advised for any future investigation with this combination in regards to toxicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No